CLINICAL TRIAL: NCT04950907
Title: A Randomized Controlled Study of Single Port Tubeless VATS for the Evaluation of Qualified Rate of Biopsy for Second-generation Tibial Specimens in Patients With Advanced NSCLC
Brief Title: Uniportal Tubeless VATS for the Evaluation of Biopsy for Second-generation Sequencing in Patients With Advanced NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jianxing He (Other)
Responsible Party: Sponsor-Investigator, Jianxing He, Prof., The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20210301
Record Dates: First submitted 2021-06-14; First posted 2021-07-06 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: NSCLC; Biopsy Technique; VATS; CT Guided Puncture Biopsy; NGS
Keywords: NSCLC; biopsy technique; VATS; CT guided puncture biopsy; NGS
MeSH Terms: interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment (Experimental): Uniportal VATS biopsy
  Interventions: Diagnostic Test: vats
- control (Active Comparator): CT-guided fine needle biopsy
  Interventions: Diagnostic Test: CT-guided fine needle biopsy

INTERVENTIONS:
Diagnostic Test: vats — Use uniportal tubeless VATS to obtain the biopsy
  Arms: treatment
Diagnostic Test: CT-guided fine needle biopsy — Use CT-guided fine needle to obtain the biopsy
  Arms: control

SUMMARY:
The study is a single-center, prospective, open-label randomized controlled study. This study evaluates the eligibility rate of different biopsy methods (tubeless tubeless VATS vs. CT guided fine needle aspiration) for the detection of molecular genetic characteristics of peripheral NSCLC next-generation sequencing, and its main purpose is to evaluate the use of tumor gene profiling (NGS) The best biopsy technique, the First Affiliated Hospital of Guangzhou Medical University is the research center. It is expected to be completed between 2021-3-1 and 2023-3-1.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent is obtained
* Assessed by more than 2 surgeons, patients whose lesions can be achieved by tubeless single-port thoracoscopic surgical biopsy

Exclusion Criteria:

* History of other malignant tumors.
* The general condition is not suitable for puncture, bronchoscopy, or surgery (such as cardiopulmonary dysfunction, high risk of bleeding, allergy to anesthetics, confusion, inability to exercise, etc.)
* History of lung surgery, tuberculosis and coal mine work experience, etc. may cause severe chest adhesions; other situations that conflict with the biopsy process

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2023-06-26 (Estimated); Study Completion 2024-06-26 (Estimated)

PRIMARY OUTCOMES:
Qualified Rate of Biopsy for Second-generation Tibial Specimens | up to 2 years
  Different biopsy methods (single-port tubeless VATS biopsy vs CT-guided fine-needle aspiration biopsy) are used to evaluate the qualification rate of samples obtained for NGS testing

SECONDARY OUTCOMES:
Progression Free Survival | up to 2 years
  Progression Free Survival of patients under different biopsy methods
Overall Survival | up to 2 years
  Overall Survival of patients under different biopsy methods
Tumor Content Size | up to 2 years
  Tumor Content of patients under different biopsy methods
Gene Mutation Rate | up to 2 years
  Gene Mutation Rate of patients under different biopsy methods
Drug sensitive mutation detection rate | up to 2 years
  Drug sensitive mutation detection rate of patients under different biopsy methods
Detection of PD-L1 expression | up to 2 years
  Detection of PD-L1 expression of patients under different biopsy methods
TMB detection situation | up to 2 years
  TMB detection situation of patients under different biopsy methods
Correlation between tumor cell content and detection rate of sensitive mutations | up to 2 years
Perioperative complications | up to 2 years
Postoperative patient experience score | up to 2 years
Usage rate of targeted drug | up to 2 years
Success rate of enrollment | up to 2 years
Postoperative MRD detection | up to 2 years